CLINICAL TRIAL: NCT00026910
Title: Analysis of Molecular Markers of Drug Resistance in Tumor Biopsies From Previously Untreated Aggressive Non-Hodgkin's Lymphoma
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980136; 98-C-0136
Record Dates: First submitted 2001-11-14; First posted 2001-11-15 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-05

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: Cell-Cycle; Apoptosis; Molecular Prognosis
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

SUMMARY:
Although the cause(s) of clinical drug resistance in non-Hodgkin's lymphomas (NHL) are unknown, in vitro studies suggest that abnormalities of the cell cycle and mechanisms of apoptosis may play an important role. Clinical studies have now shown that p53, bcl-2 and tumor proliferation all have significant effects on clinical drug resistance. To further investigate the role of genes that control the cell cycle and apoptosis, we wish to correlate the expression of multiple molecular targets [including but not restricted to bcl-2, BAX, bcl-6, MIB-1, p53, p21, p27, p16, cyclin D(1), cyclin A, cyclin E, mdm-2, cpp 32, mcl-1, EBER-1, ALK, and a panel of B, T and other cell lineage markers], involving these pathways, with clinical outcome following treatment with combination chemotherapy. All clinical data and tissue samples for this study will come from patients who have been previously enrolled on two protocols for the initial treatment of aggressive lymphomas. No new patients will be enrolled for this study.

DETAILED DESCRIPTION:
Although the cause(s) of clinical drug resistance in non-Hodgkin's lymphomas (NHL) are unknown, in vitro studies suggest that abnormalities of the cell cycle and mechanisms of apoptosis may play an important role. Clinical studies have now shown that p53, bcl-2 and tumor proliferation all have significant effects on clinical drug resistance. To further investigate the role of genes that control the cell cycle and apoptosis, we wish to correlate the expression of multiple molecular targets using immunohistochemistry and cDNA microarray expression profiling (including but not restricted to bcl-2, BAX, bcl-6, MIB-1, p53, p21, p27, p16, cyclin D1, cyclin A, cyclin E, mdm-2, cpp 32, mcl-1, EBER-1, ALK, and a panel of B, T and other cell lineage markers), involving these pathways, with clinical outcome following treatment with combination chemotherapy. All clinical data and tissue samples for this study will come from patients who have been previously enrolled on two protocols for the initial treatment of aggressive lymphomas. No new patients will be enrolled for this study.

ELIGIBILITY:
Prior enrollment on the clinical trial of ProMACE-CytaBOM versus ProMACE-MOPP (81-C-0166) or Short Course ProMACE-CytaBOM (87-C-0180) for the treatment of previously untreated aggressive lymphomas.

Informed consent for participation in the above clinical trials.

Adequate biopsy material from initial biopsy and/or biopsies at relapse of disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 1998-07; Study Completion 2002-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Harris CC, Hollstein M. Clinical implications of the p53 tumor-suppressor gene. N Engl J Med. 1993 Oct 28;329(18):1318-27. doi: 10.1056/NEJM199310283291807. No abstract available. PMID 8413413
- [Background] Wilson WH, Teruya-Feldstein J, Fest T, Harris C, Steinberg SM, Jaffe ES, Raffeld M. Relationship of p53, bcl-2, and tumor proliferation to clinical drug resistance in non-Hodgkin's lymphomas. Blood. 1997 Jan 15;89(2):601-9. PMID 9002964
- [Background] Sachs L, Lotem J. Control of programmed cell death in normal and leukemic cells: new implications for therapy. Blood. 1993 Jul 1;82(1):15-21. PMID 8324219